CLINICAL TRIAL: NCT00166478
Title: A Prospective Controlled Phase II Study of Preoperative Exisulind Therapy Initiated Prior to Radical Prostatectomy: Effect on Apoptosis
Brief Title: Exisulind Prior to Radical Prostatectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2297-01; N01-CN-75017
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Drug: Exisulind Therapy

SUMMARY:
This trial will compare no treatment to exisulind therapy. Patients enrolled on the treatment arm will begin treatment 4 weeks prior to the scheduled date of surgical removal of the prostate and will take 375 mg by mouth daily for the 4 weeks prior to radical prostatectomy. Participants will be followed for total of 2 months from the time of starting study drug.

ELIGIBILITY:
Males 40 years of age and older with prostate cancer who are scheduled to undergo surgical removal of the prostate at Mayo Clinic Rochester, Mayo Clinic Jacksonville, or Mayo Clinic Arizona may be eligible for this protocol.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2002-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
4 week changes in apoptosis biomarkers

SECONDARY OUTCOMES:
4 week changes in surrogate endpoint biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Bradley C. Leibovich, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States